CLINICAL TRIAL: NCT06523946
Title: Using Momentary Measures to Understand Physical Activity Adoption and Maintenance Among Pacific Islanders in the United States
Brief Title: Pacific Islander Physical Activity Project
Acronym: PiPA
Status: Not yet recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Ohio State University (Other); National Tongan American Society (Unknown)
Responsible Party: Principal Investigator, Neng Wan, Associate Professor, University of Utah
Other Study IDs: R37CA276365 (NIH)
Record Dates: First submitted 2024-07-12; First posted 2024-07-29 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior | interventions — dentin sialophosphoprotein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pacific Islander (PcI) Adults: The investigators will enroll 150 sedentary Pacific Islander (PcI) adults. The investigators will first use an evidence-based physical activity (PA) program tool on all participants to stimulate their PA levels, and then study how contextual and psychosocial factors influence PA initiation and maintenance. The investigators will assess participants for 5 separate weeks during a 20-month span using real-time, field-based, state-of-the-art methodologies consisting of MotionSense (a well-validated on-body mobile sensor system), ecological momentary assessment (EMA), and the Global Positioning System (GPS).
  Interventions: Behavioral: Diabetes Prevention Program (DPP) (shortened)

INTERVENTIONS:
Behavioral: Diabetes Prevention Program (DPP) (shortened) — The investigators will adapt the protocol of the 'Ohana project. The 'Ohana protocol was developed based on CDC's Diabetes Prevention Program (DPP) curriculum and designed to fit PcI's cultural background. It includes a 8-lesson curriculum delivered in 8 weeks (shortened from the original 16-lesson, 24-week core curriculum of DPP while retaining all original foci and behavior change strategies). Specifically, the first four lessons, delivered every week, focus on getting the participants started on increasing PA and improving diet (e.g., introduction; getting started on PA and diet; utilizing goal setting; making the process fun). The second four classes will be taught every other week and will focus on how to handle various challenges involved in maintaining healthy lifestyle behaviors. The investigators will deliver the curriculum in group settings of 15 people in a separate room in the National Tongan American Society.

SUMMARY:
This proposed longitudinal study will examine the influences of neighborhood factors and momentary contextual and psychosocial factors, which the investigators call acute precipitants, on physical activity (PA) adoption and maintenance among Pacific Islanders (PcIs). Specifically, the investigators will enroll 150 sedentary PcI adults and examine their PA adoption and maintenance based on measurements at five separate weeks during a 20-month period. The investigators will use MotionSense, an innovative and proven mHealth kit developed by team members, Global Positioning System (GPS), and ecological momentary assessment to measure PA and its key determinants. Our central hypotheses are that individual and neighborhood factors are associated with PA adoption and maintenance among previously sedentary PcIs, and that psychosocial precipitants mediate these associations.

DETAILED DESCRIPTION:
Pacific Islanders (PcIs), one of the fastest growing racial/ethnic groups in the United States, bear the highest obesity rate among all racial/ethnic groups in the United States and suffer from a disproportionate burden of health disparities in cardiovascular diseases, diabetes, and cancers. PA is important for addressing these disparities because regular PA decreases obesity and reduces the risks of these diseases. In general, PcIs are less physically active than non-Hispanic Whites, with the majority not meeting nationally-recommended PA levels. However, few studies have investigated the underlying mechanism(s) of PA behavior change for PcIs. Recent research highlighted the importance of contextual social and built environments on PA participation among racial/ethnic minorities and the necessity of understanding psychosocial pathways to PA behaviors. However, research in this area has been significantly limited by the lack of data measured at micro timescales (e.g., across minutes, hours, or days) that can capture the dynamic interactions between contextual factors and PA behavior. The paucity of research on PA behaviors among PcIs and the lack of micro timescale data for understanding PA mechanisms have hampered the search for effective policies and interventions to reduce PA-related health disparities for this high-risk population.

Our long-term goal is to use mobile Health (mHealth) technologies to help PcIs increase their PA levels and thereby to reduce their health disparities. This proposed longitudinal study will examine the influences of neighborhood factors and momentary contextual and psychosocial factors, which the investigators call acute precipitants, on PA adoption and maintenance among PcIs. Specifically, the investigators will enroll 150 sedentary PcI adults and examine their PA adoption and maintenance based on measurements at five separate weeks during a 20-month period. The investigators will use MotionSense, an innovative and proven mHealth kit developed by team members, GPS, and ecological momentary assessment to measure PA and its key determinants. An innovation of this mHealth system is that it can continuously measure PA and contextual and psychosocial acute precipitants in natural environments, therefore providing the much-needed micro timescale data for studying the dynamic nature of PA behavioral change. Our preliminary studies have confirmed the feasibility of using this system to measure PA and PA correlates. Our multidisciplinary team has expertise in PA behavior analysis, PA intervention, mHealth technologies, geographical analysis, and health psychology.

Our central hypotheses are that individual and neighborhood factors are associated with PA adoption and maintenance among previously sedentary PcIs, and that psychosocial precipitants mediate these associations. The investigators have designed the following two aims to test these central hypotheses.

Aim 1: To examine the influences of neighborhood factors on PA adoption and maintenance among sedentary PcI adults. The investigators hypothesize that lower levels of PA adoption and maintenance are associated with disadvantageous neighborhood factors (e.g., lack of access to PA facilities, higher levels of poverty, lower social cohesion) after controlling for individual-level factors. The investigators will first define PA adoption and maintenance based on the change of PA level across the five measurement weeks for each participant, and then link them to neighborhood factors using linear mixed effects models.

Aim 2: To determine the dynamic relationships between contextual and psychosocial acute precipitants and PA.

2.a. The investigators hypothesize that lower frequency and duration of PA are associated with disadvantageous acute precipitants (e.g., decreased access to PA facilities, increased negative affect, and decreased self-efficacy); and the associations vary between stages of PA adoption and maintenance. The investigators will use the micro timescale data measured by our mHealth system to construct PA indicators and acute precipitants. Then, an innovative dynamic prediction model will be used to investigate their temporal, dynamic associations.

2.b. The investigators hypothesize that psychosocial acute precipitants (e.g., self-efficacy, negative affect) mediate the influence of contextual acute precipitants (e.g., access to PA resources) on PA, should the investigators find any significant associations between the latter two.

This is an observational study (rather than an interventional study) that contains a physical activity intervention. The primary goal is not to evaluate the effectiveness of the PA intervention in increasing PA levels, but how neighborhood and contextual factors influence PA adoption and maintenance. The investigators use the PA intervention to stimulate PA engagement for all participants so that the investigators can observe their PA behavior change in a real-world setting.

Since the purpose of the study is not to evaluate the effectiveness of the intervention, it does not fulfill the third criterion of the NIH definition of clinical trials and should be considered an observational study.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years of age or older (because children and adolescents are different from adults in terms of PA level, PA mechanisms, psychosocial factors, and measurement accuracy);
* being Tongan American (TA); being currently sedentary which is defined as self-reported PA less than 3 days/week for less than 20 minutes/day over the last 6 month;
* no underlying functional impairment;
* valid home address;
* functioning telephone number;
* can speak, read, and write in English;
* marginal or adequate health literacy.

Exclusion Criteria:

* currently in a physical activity program or participated in a physical activity program in the past year;
* have a pacemaker or implanted cardiac device;
* have any dietary/exercise restrictions or limitations, and/or co-morbid conditions that would have precluded them from fully participating in the study;
* physically unable to wear equipment and provide a good reading or use a smartphone;
* pregnancy or lactation;
* with active diagnoses of major depression, cognitive impairment (of any etiology), or any functional impairment; or any uncontrolled medical or psychiatric problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This longitudinal cohort study will enroll 150 sedentary Tongan American (TA) adults (equally split between male and female) in Utah. Utah has the highest per-capita percentage of PcIs among the continental states, with a PcI population of 38,000 in 2014. TAs are the largest PcI group in Utah, accounting for 38% of the total PcI population. TAs primarily live in urban areas of Salt Lake and Utah counties, the two most populous counties in the state. The gender ratio is approximately 1 (i.e., 102 males to 100 females). About 7% of TAs hold a bachelor's degree, the lowest rate among all racial/ethnic groups. Although the majority live in relatively low income neighborhoods, over a quarter live in census tracts with poverty rate <5% (average median household income: $92,301), suggesting good heterogeneity in their socioeconomic status. About 27% of the TA population in Utah were foreign-born.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-08-09 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity adoption measure 1 | 5 separate weeks' data in 20 months for each participant
  Physical activity adoption will be defined in terms of change of weekly moderate-to-vigorous physical activity (MVPA) minutes during the 5 measurement weeks.
Physical activity maintenance measure 1 | 5 separate weeks' data in 20 months for each participant
  Physical activity maintenance will be defined in terms of change of weekly moderate-to-vigorous physical activity (MVPA) minutes during the 5 measurement weeks.
Physical activity adoption measure 2 | 5 separate weeks' data in 20 months for each participant
  Physical activity adoption will also be measured by a binary variable-i.e., whether the participant meets the weekly PA threshold or not.
Physical activity maintenance measure 2 | 5 separate weeks' data in 20 months for each participant
  A secondary type of physical activity maintenance would be a binary variable-i.e., whether the participant meets the weekly PA threshold or not

CONTACTS AND LOCATIONS:
Overall Officials: Neng Wan, Ph.D., Principal Investigator — Associate Professor

IPD SHARING:
Plan to Share IPD: Undecided
Data from this study will not be shared with other researchers for future studies unrelated to the study protocol. For future studies related to the study protocol, we will follow strict, IRB-approved procedures to protect participant confidentiality.